CLINICAL TRIAL: NCT07157280
Title: Quality Indicators as a Tool for Continuous Improvement Process in Clinical Obstetrics
Brief Title: Quality Indicators in Obstetrics
Acronym: QUIG
Status: Not yet recruiting | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Marcus Riemer, MD, deputy director, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: UKGEB005
Record Dates: First submitted 2025-08-22; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Quality Health Care; Quality Indicators, Health Care
Keywords: quality management; quality indicators; obstetrics; staff

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- staff in obstetrics: midwives and physicians

SUMMARY:
The study examines whether midwives and doctors are familiar with quality indicators in clinical obstetrics and whether these are used as a tool for continuous improvement process.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* staff in clinical obstetrics (midwife, physician)

Exclusion Criteria:

* nurse in clinical obstetrics
* staff in outpatient obstetrics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of midwives and doctors working in obstetrics.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Use of quality indicators | 1 year
  Number of measures taken based on the publication of quality assurance reports

IPD SHARING:
Plan to Share IPD: Undecided